CLINICAL TRIAL: NCT06269666
Title: P200TxE Diseased Eye Image Collection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Optos, PLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPT1100
Record Dates: First submitted 2024-02-13; First posted 2024-02-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Retinal Disease
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Imaging Session (Other): Various scans will be captured
  Interventions: Device: P200TxE

INTERVENTIONS:
Device: P200TxE — SLO and OCT imaging

SUMMARY:
The primary objective is to collect images on the P200TxE device in diseased eyes.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 22 years of age or older who have full legal capacity to subject on the date the informed consent is signed;
2. Subjects who can follow the instructions by the clinical staff at the clinical site;
3. Subjects who agree to participate;
4. Subjects who have been diagnosed with retinal pathology and/or glaucoma that affects the posterior pole region including the macula and/or optic nerve.

For glaucoma subjects:

a. Glaucoma subjects who have a history of visual field loss and RNFL or optic nerve changes.

Exclusion Criteria:

1. Subjects unable to tolerate ophthalmic imaging;
2. Subjects with ocular media not sufficiently clear to obtain acceptable images.

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of images | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Bennett and Bloom Eye Centers, Louisville, Kentucky, United States